CLINICAL TRIAL: NCT06828042
Title: A Single-center Clinical Study Evaluating the Safety and Efficacy of Universal CD19-targeting CAR-γδT Cells（QH103） in Refractory Autoimmune Diseases
Brief Title: Safety and Efficacy of Universal CD19-targeting CAR-γδT Cells in Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20250025
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erthematosus; Systemic Sclerosis (SSc); Sjogren Syndrome; ANCA Associated Vasculitis (AAV); Inflammatory Myopathies; Antiphospholipid Syndrome
MeSH Terms: conditions — Scleroderma, Systemic; Sjogren's Syndrome; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 CAR-γδ T (Experimental)
  Interventions: Biological: anti-CD19 CAR T cell therapy

INTERVENTIONS:
Biological: anti-CD19 CAR T cell therapy — anti-CD19 CAR-γδ T cell therapy

SUMMARY:
Autoimmune diseases refer to a common category of diseases caused by the immune system reacting to self-antigens, leading to tissue damage. Autoimmune diseases encompass a wide variety of conditions, such as systemic lupus erythematosus（SLE）, Sjögren's syndrome (SS), systemic sclerosis (SSc), inflammatory myopathies (IM), ANCA-associated vasculitis (AAV), and antiphospholipid syndrome (APS). They affect the quality of life, while in severe cases, they can be life-threatening. Additionally, they impose a heavy economic burden on society. Current treatments for autoimmune diseases include glucocorticoid, immunosuppressants, and biologics. B cell-driven humoral immune abnormalities are a central pathogenic mechanism in many autoimmune diseases. When autoreactive B cells are excessively activated, they produce large amounts of autoantibodies and immune complexes. These antibodies and immune complexes can cause damage to various tissues and organs, leading to the development of multiple autoimmune diseases. Therefore, targeting B cells to treat autoimmune diseases is an attractive therapeutic strategy.

Chimeric Antigen Receptor (CAR)-T cells targeting the B cell surface molecule CD19 have achieved significant clinical progress in acute lymphoblastic leukemia and B cell non-Hodgkin lymphoma, with several CD19 CAR-T therapies approved for marketing worldwide. Increasingly, clinical studies are exploring the use of CD19 CAR-T cells for the treatment of autoimmune diseases, and their therapeutic efficacy has been demonstrated.

In this study, the investigators used γδ T cells as carrier cells to investigate the safety and efficacy of universal CAR-γδ T cells in the treatment of autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

Common Inclusion Criteria:

1. Age between 18-80 years (inclusive), male or female.
2. Positive expression of CD19 on peripheral blood B cells by flow cytometry.
3. Diagnosed with refractory autoimmune disease, defined as: Ineffectiveness of conventional treatment for more than 6 months, or Disease activity recurrence after remission. Definition of conventional treatment: Use of glucocorticoids and any of the following immunosuppressants or biologics: cyclophosphamide, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, rituximab, belimumab, telitacicept, etc.
4. Currently receiving one or more standard therapies at a stable dose, including glucocorticoids, antimalarials, immunosuppressants, or biologics. If the subject is receiving glucocorticoids, the following conditions must be met: During screening and the screening period, the maximum dose of glucocorticoids is 30 mg/day prednisone (or an equivalent dose). The glucocorticoid dose must remain stable for ≥7 days before screening, and during the screening period, the dose adjustment must not exceed >5 mg/day prednisone (or an equivalent dose). If the subject is receiving antimalarials and/or conventional immunosuppressants: The treatment must have started ≥12 weeks before screening. The medication dose must remain stable for ≥8 weeks before screening and throughout the screening period. Before cell infusion, other immunosuppressants (excluding hydroxychloroquine), including belimumab, telitacicept, CD20 monoclonal antibodies, or other biologic immunosuppressants, must be discontinued for at least 5 half-lives.
5. Female participants of childbearing potential and male participants with female partners of childbearing potential must use medically approved contraceptive methods or practice abstinence during the study treatment period and for at least 6 months after the study. Female participants of childbearing potential must have a negative serum HCG test within 7 days before enrollment and must not be breastfeeding.
6. Willing to participate in the trial and sign the informed consent form.

Disease-Specific Inclusion Criteria:

1. Systemic Lupus Erythematosus (SLE):

   * Meets the 2019 EULAR/ACR classification criteria for SLE.
   * ANA titer ≥1:80, or positive for anti-dsDNA and/or anti-Sm antibodies.
   * Disease activity score (SLEDAI-2000) ≥8.
2. Sjögren's Syndrome:

   * Meets the 2002 AECG criteria or the 2016 ACR/EULAR classification criteria for primary Sjögren's syndrome.
   * Disease activity score (ESSDAI) ≥5.
   * Positive for anti-SSA/Ro antibodies.
3. Systemic Sclerosis (SSc):

   * Meets the 2013 EULAR/ACR classification criteria for systemic sclerosis.
   * Classified by Leroy and Medsger as limited or diffuse cutaneous subsets.
   * At screening, mRSS >10; and/or active interstitial lung disease (ILD), defined as: High-resolution computed tomography (HRCT) showing ground-glass opacities. Pulmonary function tests (FVC or DLCO) <70% of predicted values.
4. Idiopathic Inflammatory Myopathies (IIM):

   * Meets the 2017 EULAR/ACR classification criteria for inflammatory myopathies (including dermatomyositis, polymyositis, antisynthetase syndrome, and necrotizing myopathy).
   * For patients with muscle involvement: a. MMT-8 score <142 and at least two abnormal findings among the following core measures: PhGA or PtGA scores ≥2. Extramuscular disease activity score ≥2. HAQ total score ≥0.25. Muscle enzyme levels ≥1.5 times the upper normal limit. b. Alternatively, MMT-8 ≥142 but with active ILD (HRCT showing ground-glass opacities).
   * Positive for myositis-specific antibodies.
5. ANCA-Associated Vasculitis (AAV):

   * Meets the 2022 ACR/EULAR diagnostic criteria for ANCA-associated vasculitis, including microscopic polyangiitis, granulomatosis with polyangiitis, or eosinophilic granulomatosis with polyangiitis.
   * Positive for ANCA antibodies (current or historical).
   * Birmingham Vasculitis Activity Score (BVAS) ≥15 (out of 63), indicating active vasculitis.
6. Refractory Antiphospholipid Syndrome (APS):

   * Meets the 2023 ACR/EULAR diagnostic criteria for antiphospholipid syndrome.
   * Positive for medium-to-high titers of antiphospholipid antibodies (LA, anti-β2-GP1, or ACL IgG/IgM), with at least two positive results within 3 months.
   * Definition of refractory APS: Disease remains active or relapses after remission, despite 6 months of conventional therapy, including: Anticoagulants (warfarin or standard treatment with vitamin K antagonists maintaining target INR) or low-molecular-weight heparin at standard doses. Glucocorticoids and/or immunosuppressants.
   * Catastrophic APS (CAPS): Must meet all four criteria: a. Involvement of three or more organs, systems, and/or tissues. b. Symptoms occurring within one week. c. Histological evidence of small vessel occlusion in at least one organ or tissue. d. Positive for antiphospholipid antibodies (aPL).

Note: Meeting either criterion 3 or 4 is sufficient. Patients with thrombocytopenia may not require anticoagulant therapy.

Exclusion Criteria:

1. History of severe drug allergies or allergic constitution.
2. Presence or suspicion of uncontrolled or treatment-requiring fungal, bacterial, viral, or other infections.
3. Central nervous system (CNS) diseases caused by autoimmune or non-autoimmune conditions, including epilepsy, psychiatric disorders, organic brain syndrome, cerebrovascular accidents, encephalitis, or CNS vasculitis.
4. Dysfunction of major organs not meeting the following criteria (exceptions allowed if abnormalities are caused by autoimmune disease): a. Bone marrow function: White blood cell count ≥3×10⁹/L. Neutrophil count ≥1×10⁹/L (without GSF treatment within 2 weeks prior to testing). Hemoglobin ≥60 g/L. Platelet count ≥50×10⁹/L. b. Liver function: ALT ≤3×ULN (exceptions for ALT elevation caused by inflammatory myopathy). AST ≤3×ULN (exceptions for AST elevation caused by inflammatory myopathy). IBIL ≤1.5×ULN (exceptions for Gilbert's syndrome). Total bilirubin ≤3.0×ULN. c. Renal function: Creatinine clearance (CrCl) ≥30 mL/min (calculated using the Cockcroft/Gault formula, exceptions for acute CrCl decline caused by the disease itself). d. Coagulation function: International normalized ratio (INR) ≤1.5×ULN. Prothrombin time (PT) ≤1.5×ULN. e. Cardiac function: Stable hemodynamics.
5. Subjects with congenital immunoglobulin deficiencies.
6. History of malignancy within the past five years.
7. Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood HBV DNA levels exceeding the detection limit; positive hepatitis C virus (HCV) antibodies with detectable HCV RNA in peripheral blood; positive HIV antibodies; or positive syphilis test results.
8. Subjects with psychiatric disorders or severe cognitive impairment.
9. Participation in other clinical trials within 3 months prior to enrollment.
10. Previous treatment with CAR-T therapy.
11. History of severe adverse reactions to cyclophosphamide or fludarabine.
12. Any other reason that the investigator determine that subjects cannot be included in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of QH103（anti-CD19 CAR-γδT cells） | 0-Month 12
  Incidence of Treatment-Emergent Adverse Events (AEs) in this study. AEs are defined as any adverse medical events occurring from the initiation of lymphodepleting chemotherapy to 12 months after the completion of QH103 cell infusion. The incidence, duration, severity, and management of all adverse events occurring after the participants' enrollment will be recorded and evaluated.Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Graft-versus-host disease (GVHD) will be graded based on the criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE, v5.0).
Maximum tolerated dose of CD19 CAR-γδT cells | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2000) score | Month 3, 6, 9, and 12
  The change from baseline in the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2000) score at Month 3, 6, 9, and 12.
SRI-4 response | month 3, 6, 9, and 12
  SLE patients who met all three of the following conditions at month3,6,9, and 12 after infusion, achieve SRI-4 response:
  1. The SLEDAI-2K rating dropped by at least 4 points
  2. No deterioration in PGA scores on a 3-point scale (deterioration is defined as an increase of ≥0.3 points from baseline score)
  3. No new manifestations of organ system involvement (new system involvement is defined as one or more new symptoms of BILAG grade A or two or more symptoms of BILAG B)
Sjögren's Tool for Assessing Response (STAR) score | Month 3, 6, 9, and 12.
  The changes from baseline in the Sjögren's Tool for Assessing Response (STAR) score at Month 3, 6, 9, and 12.
EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) | Month 3, 6, 9, and 12
  The changes from baseline in the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) at Month 3, 6, 9, and 12.
EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) | Month 3, 6, 9, and 12
  The changes from baseline in the EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) at Month 3, 6, 9, and 12.
Systemic Sclerosis Combined Response Index (CRISS) response | Month 3, 6, 9, and 12
  Patients achieve Systemic Sclerosis Combined Response Index (CRISS) response Month 3, 6, 9, and 12. A responder meets all of the following criteria; otherwise, they are classified as a non-responder.
  1. Improvement in at least two aspects (≥ 5% increase in ppFVC and/or ≥ 25% decrease in mRSS, HAQ-DI, PtGA, or PhGA);
  2. Worsening in no more than one aspect (≥ 5% decrease in ppFVC and/or ≥ 25% increase in mRSS, HAQ-DI, PtGA, or PhGA);
  3. No significant new SSc-related manifestations.
Modified Rodnan Skin Score (mRSS) | Month 3, 6, 9, and 12
  The changes from baseline in the modified Rodnan Skin Score (mRSS) at Month 3, 6, 9, and 12.
Total Improvement Score (TIS) | Month 3, 6, 9, and 12
  For IM patients with a baseline MMT-8 score <142, the changes from baseline in Total Improvement Score (TIS) based on the Myositis Response Criteria, which includes changes in the physician's global assessment, the patient's global assessment, the health assessment questionnaire (SF-36), manual muscle testing (MMT-8), muscle enzymes, and extramuscular disease activity at month 3, 6, 9, and 12.
Improvement in interstitial lung disease | Month 3, 6, 9, and 12
  For IM patients with a baseline MMT-8 score ≥142, the assessment of improvement in interstitial lung disease, defined as an increase of ≥10% in forced vital capacity (FVC) or diffusing capacity for carbon monoxide (DLCO) compared to baseline at Month 3, 6, 9, and 12.
Vasculitis disease activity assessment (BVAS score) | Month 3, 6, 9, and 12
  The changes from baseline in vasculitis disease activity assessment (BVAS score) for patients with AAV at Month 3, 6, 9, and 12
Vasculitis Damage Index (VDI) | Month 3, 6, 9, and 12
  The changes from baseline in the Vasculitis Damage Index (VDI) for AAV patients at Month 3, 6, 9, and 12.
Newly developed, imaging-confirmed thrombosis in APS patients | Month 3, 6, 9, and 12
  Newly developed, imaging-confirmed thrombosis in APS patients at Month 3, 6, 9, and 12.
Platelet count for APS patients | Month 3, 6, 9, and 12
  The changes from baseline in platelet count for APS patients at Month 3, 6, 9, and 12.
PD parameters | 0-Month 3
  The Changes from baseline of level IL-6 in peripheral blood after infusion of QH103
PK-Tmax | 0-Month 3
  Time to peak in CAR-T cell count in peripheral blood after infusion of QH103.
PK-Cmax | 0-Month 3
  Peak concentration (Cmax) in the CAR-T cell count in peripheral blood after infusion of QH103
PK-AUC | 0-Month 3
  Area under the concentration-time curve of CAR-T cell count in peripheral blood after infusion of QH103 from 0 to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
No decision has been made regarding the issue